CLINICAL TRIAL: NCT03793881
Title: Effectiveness of a Nutritional Strategy for Blood Pressure Control in Patients With Hypertension Users of a Public Health System: NUPRESS Study
Brief Title: Nutritional Strategy for Blood Pressure Control in Patients With Hypertension (NUPRESS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NUPRESS
Record Dates: First submitted 2019-01-03; First posted 2019-01-04 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2022-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutritional Strategy (Experimental): Nutritional counseling based on the quality of the diet, the Food Guide for the Brazilian Population and concepts of mindfulness and mindful eating; dietary guidance based on feasible goals built together (patient and nutritionist).
  Interventions: Behavioral: Nutritional Strategy
- Dietary Prescription (Active Comparator): Individualized dietary prescription according to the guidelines of the Brazilian Society of Cardiology.
  Interventions: Behavioral: Dietary Prescription

INTERVENTIONS:
Behavioral: Nutritional Strategy — Counseling based on dietary goals and mindfulness techniques.
  Arms: Nutritional Strategy
Behavioral: Dietary Prescription — Dietary prescription according to guidelines.
  Arms: Dietary Prescription

SUMMARY:
Adherence to a healthy dietary pattern is part of the self-care of patients with hypertension, and may contribute substantially to therapeutic target goals as well as to a better quality of life. However, not all nutritional recommendations aimed at these patients are easily applicable in clinical practice. The primary objective of the study is to evaluate the effectiveness of a nutritional strategy for blood pressure control in patients with hypertension users of a Public Health System after 6 months of follow-up. As secondary objectives, we will evaluate the impact of the proposed strategy on self-care and on the quality of life of the patients. In this multicenter open-label randomized trial, 408 patients ≥21 years old with hypertension, systolic blood pressure (SBP) ≥140mmHg at the moment of the screening and who have not received or received nutritional counseling for at least 06 months will be enrolled. Patients allocated to the control group will receive individualized dietary prescription according to the guidelines of the Brazilian Society of Cardiology. Nutritional counseling in the intervention group will be performed based on the quality of the diet, the Food Guide for the Brazilian Population and concepts of mindfulness and mindful eating; all dietary guidance will be based on feasible goals built together (patient and nutritionist), and no diet will be prescribed for intervention group. In both groups, patients will receive automatic monitors for residential self-monitoring blood pressure. On-site follow-up visits will be carried out at 30, 60, 90, and 180 days (final consultation). At 120 and 150 days, participants in the intervention group will receive motivational messages via e-mail or SMS (for these patients, consultation of 30 days will be a group meeting). Laboratory tests (lipid and glycemic profile, serum creatinine, serum sodium, urinary sodium, serum potassium, urinary potassium and albuminuria) will be performed at baseline and 180 days; anthropometric indexes and diastolic blood pressure (DBP) will be also evaluated.

ELIGIBILITY:
Inclusion Criteria: ≥21 years old with medical diagnosis of hypertension, systolic blood pressure (SBP) ≥140 mmHg at the moment of the screening and who have not received or received nutritional counseling for at least 06 months.

Exclusion Criteria:

* Diagnosis of resistant and/or secondary hypertension;
* Severe neuropathy;
* Chronic kidney disease;
* Active cancer or life expectancy <6 months;
* Chemical dependence or use of antipsychotic drugs;
* Autoimmune disease or chronic use of steroids;
* Pregnancy and lactation;
* Acute coronary syndrome in the last 60 days;
* Severe or unstable heart failure;
* Wheelchair users;
* Extreme obesity (body mass index [BMI] ≥40kg / m²);
* Cognitive, neurological or psychiatric condition that prevents participation in the study;
* Participation in other clinical trials.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2021-07-22 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
SBP | 6 months
  Systolic blood pressure, in mmHg
BPC | 6 months
  Blood pressure control, defined as either having systolic blood pressure (SBP) > 140 mmHg at baseline and achieving SBP ≤ 140 mmHg after follow-up or having SBP ≤ 140 mmHg at baseline and reducing anti-hypertensive drugs after follow-up.

SECONDARY OUTCOMES:
DBP | 6 months
  Diastolic blood pressure, in mmHg
HbA1C | 6 months
  Glycated hemoglobin, in %
FG | 6 months
  Fasting glucose, in mg/dL
BW | 6 months
  Body weight, in kg
WC | 6 months
  Waist circumference, in cm
BMI | 6 months
  Body mass index, in kg/m2; it will be defined according to the mathematical formula (BW/height*height)
TC | 6 months
  Total cholesterol, in mg/dL
LDL-c | 6 months
  LDL cholesterol, in mg/dL; it will be defined according to the Martin´s mathematical formula
HDL-c | 6 months
  HDL cholesterol, in mg/dL
TG | 6 months
  Serum triglycerides, in mg/dL
VLDL-c | 6 months
  VLDL cholesterol, in mg/dL; it will be obtained according to the mathematical formula TG/5
NHDL | 6 months
  Non-HDL cholesterol, in mg/dL; it will be obtained according to the mathematical formula TC-HDL-c
Castelli Index I | 6 months
  Castelli Index I, in mg/dL; it will be obtained according to the mathematical formula TC/HDL-c
Castelli Index II | 6 months
  Castelli Index II, in mg/dL; it will be obtained according to the mathematical formula LDL-c/HDL-c
Cr | 6 months
  Creatinine, in mg/dL
GFR | 6 months
  Glomerular filtration rate, in ml/min/1.73m2
Sodium (s) | 6 months
  Serum sodium, in mEq/L
Sodium (u) | 6 months
  Urinary sodium, in mEq/L
Potassium (s) | 6 months
  Serum potassium, in mEq/L
Potassium (u) | 6 months
  Urinary potassium, in mEq/L
ALB | 6 months
  Albuminuria, in mg/g
DQ | 6 months
  Diet quality, assessed by the modified Alternative Healthy Eating Index (mAHEI)
MINICHAL | 6 months
  Quality of life evaluated by the Brazilian version of the Mini-cuestionario de calidad de vida en la hipertensión arterial. In this tool, ten items are related to the "mental status" domain and six items to "somatic manifestations". Questions refer to the past seven days. The score scale is a likert-type scale with four possible answers (0=absolutely no; 1=yes, a little; 2=yes, fairly; 3=yes, a lot). The points range from 0 (best health level) to 30 (worst health level) for the "mental status" dimension, and from 0 (best health level) to 18 (worst health level) for the "somatic manifestations" dimension.
SHIQ | 6 months
  Self-care evaluated by the Brazilian version of the Self-care of Hypertension Inventory Questionaire. This tool includes 23 items divided across 3 scales: Self-care Maintenance (11 items), Self-care Management (6 items), and Self-care Confidence (6 items). Items in the instrument are scored on a Likert-type scale. In the Self-care Maintenance domain, scores range from 1 to 5 (''never'' to ''always''). In the Self-care Management domain, 2 items range from 0 to 5 to capture a fully negative response, and other item options are scored 1 to 5. The remaining items are scored from 1 to 5 (''not likely'' to ''very likely''). In the self-care confidence scale, items are scored from 1 to 5. Scores are calculated for each scale individually. Each scale is standardized to range from 0 to 100. Self-care is considered adequate if the score is 70 or greater.

OTHER OUTCOMES:
TT | 6 months
  Therapeutic targets, defined as the proportion of participants who reached the following therapeutic targets: SBP/DBP < 140/90 mmHg; fasting glucose <100 mg/dL; LDL-c <100 mg/dL; BMI < 25 kg/m2 or weight loss > 5%
AHD | 6 months
  Anti-hypertensive drugs, defined as the type and proportion of anti-hypertensive drugs used

CONTACTS AND LOCATIONS:
Overall Officials: Aline Marcadenti, PhD, Principal Investigator — Hospital do Coracao
Locations (8):
- Brazil (8):
  - Universidade de Fortaleza, Fortaleza
  - Hospital de Clínicas de Goiás - Universidade Federal de Goiás, Goiânia
  - Universidade Federal de Tocantins, Palmas
  - Instituto de Cardiologia do Rio Grande do Sul, Porto Alegre
  - Pontifícia Universidade Católica do Rio Grande do Sul, Porto Alegre
  - Universidade de São Paulo, Ribeirão Preto
  - Hospital do Coracao, São Paulo
  - Hospital Comunitário São Peregrino Lazziozi, Veranópolis

IPD SHARING:
Plan to Share IPD: Yes
Data and materials will be available upon reasonable request for the corresponding author, after filling a specific form provided by IP-HCor and considering institutional data sharing politics.
Time Frame: Data will be available after main paper publication.